CLINICAL TRIAL: NCT06919523
Title: Clinical Study to Evaluate the Efficacy and Safety of Dapagliflozin in Patients With Refractory Cirrhotic Ascites
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha Mansour, Associate professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-NM
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Refractory Ascites
Keywords: Refractory ascites; Dapagliflozin
MeSH Terms: conditions — Ascites | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin group (Experimental)
  Interventions: Drug: Dapagliflozin 5mg
- Standard care only group (Active Comparator)
  Interventions: Drug: Standard care treatment

INTERVENTIONS:
Drug: Dapagliflozin 5mg — Dapagliflozin 5m orally once daily for 3 months plus standard care (diuretics and Large volume paracentesis)
  Arms: Dapagliflozin group
Drug: Standard care treatment — Diuretics and Large volume paracentesis as indicated
  Arms: Standard care only group

SUMMARY:
The aim of this clinical trial is to evaluate the safety and efficacy of low dose dapagliflozin use along with standard care versus the standard care alone in improving the clinical outcomes of patients with cirrhotic refractory ascites. The main question it aims to answer is the difference in ascites control between the two groups at the end of treatment defined as:

Complete response: Disappearance of ascites. Partial response: Presence of ascites not requiring LVP. No response: Presence of ascites requiring LVP. Researchers will compare intervention group receiving dapagliflozin 5m once daily for 3 months along with standard care versus standard care group to evaluate the effectiveness and safety of dapagliflozin in refractory ascites patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years diagnosed with decompensated liver cirrhosis complicated with ascites grade 2.
* Refractory ascites defined as one of the following:

  1. Ascites cannot be mobilized despite adherence to low sodium diet of ≤88 mmol/day for ≥1 week and maximum diuretic treatment dose (spironolactone 400 mg/day or furosemide (160 mg/day).
  2. Recurrence can't be prevented by medical therapy, Re-appearance of grade 2 or moderate ascites with moderate symmetrical abdominal distention, or grade 3 with massive ascites with marked abdominal distention within 4 weeks of initial mobilization.

Exclusion Criteria:

* Presenting blood pressure below 90/60 or history of hypotension requires vasopressor treatment.
* History of recurrent urinary tract infections, defined by the occurrence of 2 or more acute UTIs within months or 3 within a year.
* History of hypersensitivity to SGLT2 inhibitors.
* History of diabetic ketoacidosis or presence of risk factors for DKA (i.e alcohol consumption, type 1 diabetes).
* Pregnant or lactating women.
* History of recurrent episodes of hypoglycemia defined as plasma glucose concentration <70mg/dL.
* Severe renal dysfunction defined as, eGFR <20 ml/min/1.73m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Difference in ascites control between the two groups at the end of treatment | 3 months
  Complete response: Disappearance of ascites. Partial response: Presence of ascites not requiring LVP. No response: Presence of ascites requiring LVP.